CLINICAL TRIAL: NCT06612268
Title: A Global Phase 3, Randomised, Double-blind and Placebo-controlled Study Evaluating the Efficacy and Safety of Etavopivat in Adolescents and Adults With Sickle Cell Disease
Brief Title: A Study to Evaluate How Well Etavopivat Works in People With Sickle Cell Disease
Acronym: Hibiscus 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7535-7807; U1111-1298-3431 (Other: World Health Organisation (WHO)); 2023-509175-16 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etavopivat (Experimental): Participants will be randomised to receive oral dose of Etavopivat.
  Interventions: Drug: Etavopivat
- Placebo (Placebo Comparator): Participants will be randomised to receive oral dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etavopivat — Etavopivat will be administered orally.
  Arms: Etavopivat
Drug: Placebo — Placebo matching Etavopivat will be administered orally.
  Arms: Placebo

SUMMARY:
This study is conducted to confirm whether etavopivat works well at reducing the number of Vaso-occlusive crisis VOCs (sickle cell pain crises) caused by obstructions in blood vessels in adults and adolescents living with sickle cell disease. The study will also evaluate how well etavopivat can reduce the damage to different organs, improve your exercise tolerance and reduce fatigue in people with sickle cell disease.The participants will either get etavopivat or placebo. Which treatment the participants will get is decided by chance. Etavopivat is a new medicine and is currently being tested in other studies in addition to this one. The study will last for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 12 years or above at the time of signing the informed consent.
* Confirmed diagnosis of sickle cell disease: Documentation of sickle cell disease (SCD) genotype (HbSS, HbSβ0-thalassemia or other sickle cell syndrome variants) based on prior history of laboratory testing or screening test results from central laboratory. Molecular genotyping is not required. SCD genotype may be determined from the results of haemoglobin (Hb) electrophoresis, high-performance liquid chromatography (HPLC) or similar testing. Note that Hb electrophoresis is performed by the central laboratory at screening.
* Have 1-15 episodes of documented vaso occlusive crises (VOC) within the 12 months prior to screening. Documentation must exist in the participant's medical record prior to randomisation. Events based solely on participant recall without supporting documentation should not be counted towards eligibility.
* Hb greater than or equal to (≥) 5.0 and less than or equal to (≤) 10.0 g/dL (greater than or equal to (≥) 50 and less than or equal to (≤) 100 g/L) at screening.

Exclusion Criteria:

* More than 15 VOCs within the past 12 months prior to screening documented in the participant's medical record. Events based solely on participant recall without supporting documentation should not be counted towards eligibility.
* Use of voxelotor or similar agent within 28 days prior to starting study treatment or anticipated need for this agent during the study.
* Use of a selectin antagonist (e.g., crizanlizumab, monoclonal antibody or small molecule) within 28 days or 5 half-lives (whichever is longer) prior to starting study treatment or anticipated need for such agents during the study.
* Receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) or greater than or equal to 6 transfusion events in the previous 12 months (i.e., an average of 1 transfusion event every 60 days).
* Participants who have received an RBC transfusion for any reason within 60 days of the screening period or 60 days of the randomisation day are only eligible if HbA (adult haemoglobin) less than 10% by Hb electrophoresis is documented prior to starting study treatment.
* Receiving or use of concomitant medications that are strong inducers of CYP3A4 (cytochrome p450 3a4) within 2 weeks of starting study treatment or anticipated need for such agents during the study.
* Use of erythropoietin or other haematopoietic growth factor treatment within 28 days of starting study treatment or anticipated need for such agents during the study.
* Receipt of prior cellular-based therapy (e.g., haematopoietic cell transplant, gene modification therapy).
* Hepatic dysfunction characterized by:

  * Alanine aminotransferase (ALT) greater than 4.0 × upper limit of normal (ULN) or
  * Direct bilirubin greater than 3.0 × ULN.
* Participants who are not taking or are unable to take antimalarial prophylaxis at the time of consent and during the study if they live in areas of endemic malaria where prophylaxis is recommended.
* Severe renal dysfunction (estimated glomerular filtration rate [eGFR] at screening, calculated by the central laboratory greater than 30 mL/min/1.73 m^ 2) or on chronic dialysis.
* Travelled distance on standardized 6MWT below 100m at screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-08-27 (Estimated); Study Completion 2029-03-12 (Estimated)

PRIMARY OUTCOMES:
Number of adjudicated Vaso-occlusive crisis (VOC) events with a medical contact | Baseline (week 0) to week 52
  Measured as Count of events.

SECONDARY OUTCOMES:
Change in Haemoglobin (Hb) greater than 1 grams per decilitre (g/dL) | Baseline (week 0) to week 24
  Measured in Count of participants.
Time to onset of first adjudicated Vaso-occlusive crisis (VOC) | Baseline (week 0) to week 52
  Measured as time in days.
Change in standardised T-score on the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue 7a Scale | Baseline (week 0) to week 52
  Measured in T-score.
Change in haemoglobin (Hb) | Baseline (week 0) to week 52
  Measured in grams per decilitre (g/dL).
Change in lactate dehydrogenase (LDH) | Baseline (week 0) to week 52
  Measured in Units per litre (U/L).
Change in absolute reticulocyte count | Baseline (week 0) to week 52
  Measured as Cells x10^9/L.
Change in indirect bilirubin | Baseline (week 0) to week 52
  Measured in milligrams per decilitre (mg/dL).
Change in distance travelled during the 6-minute walking test (6MWT) | Baseline (week 0) to week 52
  Measured in Meters.
Participants achieving the threshold for clinically meaningful change (yes/no) in PROMIS fatigue scale 7a | Baseline (week 0) to week 52
  Measured as Count of participants.
Participants achieving the threshold for clinically meaningful change (yes/no) in 6MWT | Baseline (week 0) to week 52
  Measured as Count of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (162):
- United States (49):
  - Uni of Alabama at Birmingham, Birmingham, Alabama
  - Univer South Alabama Ped/Onc, Mobile, Alabama
  - Phoenix Children's Hsptl, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - UCLA Health, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - University Of California Irvine, Orange, California
  - Stanford University_Palo Alto, Palo Alto, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Clinical and Transl Res Center, Aurora, Colorado
  - Nemours/AI duPont Hosp-Chld, Wilmington, Delaware
  - Childrens National Medical Ctr, Washington D.C., District of Columbia
  - MedStar Hlth Res Institute, Washington D.C., District of Columbia
  - Memorial Healthcare, Hollywood, Florida
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Childrens Hospital of Chicago, Chicago, Illinois
  - Univer Of Illinois at Chicago, Chicago, Illinois
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital_Detroit, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University-St.Louis, St Louis, Missouri
  - Children's Nebraska, Omaha, Nebraska
  - Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - NYC Health+Hospitals, Brooklyn, New York
  - Interfaith Medical Center, Brooklyn, New York
  - Northwell Health, Mount Kisco, New York
  - Cohen Children's Medical Ctr, Queens, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Ctr, The Bronx, New York
  - Duke Comprehen Sickle Cell, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina Univ-Greenville, Greenville, North Carolina
  - Atrium Health-Wake Forest Bapt, Winston-Salem, North Carolina
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Ohio State Univ Wexner Med Ctr, Columbus, Ohio
  - Univ of OK Health Sciences Ctr, Oklahoma City, Oklahoma
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - St. Jude Children's Res Hosp, Memphis, Tennessee
  - UT Health University of Texas, Houston, Texas
  - Inova Health System, Fairfax, Virginia
  - Children's Hsptl Of The Kings, Norfolk, Virginia
  - Virginia Comm Univ Medical Ctr, Richmond, Virginia
  - Mary Bridge Children's Health, Tacoma, Washington
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales Hospital - Department of Haematology, Randwick, New South Wales
  - Monash Health, Clayton, Victoria
  - Fiona Stanley Hospital - Haemophilia and Haemostasis Centre, Murdoch, Western Australia
- Belgium (6):
  - CHU Saint-Pierre - UMC Sint-Pieter, Brussels
  - CHU - UVC Brugmann, Brussels
  - HUB - Hôpital Erasme, Brussels
  - UZ Antwerpen - UZA - Haematology, Edegem
  - UZ Antwerpen - UZA - Kinderhemato-Oncologie, Edegem
  - UZ Leuven - Kindergeneeskunde, Leuven
- Brazil (6):
  - MultiHemo - Grupo Oncoclínicas, Recife, Pernambuco
  - Hemocentro UNICAMP, Distrito de Barão Geraldo - Campinas, São Paulo
  - HC da FMUSP Hospital das Clínicas São Paulo, São Paulo, São Paulo
  - Fundação Hemocentro de Ribeirão Preto, Ribeirão Preto, São
  - Hemorio-Fundarj, Rio de Janeiro
  - Hospital Samaritano Higienópolis - Instituto de Conhecimento Ensino e Pesquisa (ICEP), São Paulo
- Canada (9):
  - Foothills Med Ctr-Univ Calgary, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - University of Alberta_Edmonton, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - LHSC - Victoria Hospital, London, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - CHUM-Hosp de Univ Montreal, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
- Colombia (8):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Clinica de la Costa, Barranquilla, Atlántico
  - Sociedad de Oncología y Hematología del Cesar SAS (SOHEC), Valledupar, Cesar Department
  - Clínica IMAT Oncomedica Auna S.A.S., Montería, Departamento de Córdoba
  - Centro de investigaciones clínicas, fudación valle del lili, Cali, Valle del Cauca Department
  - Sociedad de Oncología y Hematología del Cesar SAS (SOHEC), Antioquia
  - Centro de investigaciones clínicas, fudación valle del lili, Cali
  - Clínica IMAT Oncomedica Auna S.A.S., Montería
- France (8):
  - Ap-Hp-Hopital Avicenne, Bobigny
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Pellegrin, Bordeaux
  - Ap-Hp-Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon, Grenoble
  - Hospices Civils de Lyon-Hopital Edouard Herriot, Lyon
  - AP-HP-HOPITAL NECKER_Service d'hématologie, Paris
  - Ap-Hp-Hopital Robert Debre, Paris
  - Centre Hospitalier Universitaire de Rouen-Hopital Charles Nicolle, Rouen
- Ghana (3):
  - Kintampo Health Research Centre (KHRC), Kintampo, Bono East
  - Navrongo Health Research Centre, Navrongo, Upper East Region
  - Agogo Presbyterian Hospital, Ghana, Agogo
- Greece (5):
  - "Laiko" General Hospital of Athens, Athens
  - Childrens' Hospital of Athens "Agia Sofia", Athens
  - Hippokration Hospital, Athens
  - University General Hospital Of Ioannina, Ioannina
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
- India (14):
  - Gauhati Medical College and Hospital, Guwahati, Assam
  - All India Institute of Medical Sciences (AIIMS), Raipur, Raipur, Chhattisgarh
  - Zydus Medical College & Hospital, Dohad, Gujarat
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - SSG Hospital, Baroda, Vadodara, Gujarat
  - HOCC Haemato Oncology Care Centre, Vadodara, Gujarat
  - JSS Hospital, Mysore, Mysuru, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Arihant Multispeciality Hospital, Nagpur, Maharashtra
  - IMS and SUM Hospital, Bhubaneswar, Odisha
  - RNT Medical College, Udaipur, Rajasthan
  - NIZAM'S Institute of Medical Sciences, Hyderabad, Telangana
  - Post Graduate Institute of Child Health, Noida, Uttar Pradesh
  - All India Institute of Medical Sciences_New Dehli, New Delhi
- Italy (10):
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga - S.C.D.O. Microcitemie e malattie rare ematologiche, Orbassano, Torino
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona Policlinico GB Rossi - Borgo Roma - Centro Ricerche Cliniche Di Verona S.r.l., Verona, Veneto
  - ASST Civili di Brescia, Brescia
  - ARNAS Garibaldi Catania - Presidio Ospedaliero Garibaldi-Centro, Catania
  - Azienda Ospedaliero Universitaria Di Modena - UOC Pediatria ad indirizzo Oncoematologico, Modena
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - A.O.U. Università Studi della Campania "Luigi Vanvitelli", Naples
  - Azienda Ospedale Universita Padova, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo
- Kenya (4):
  - Gertrude's Children's Hospital, Nairobi, Nairobi County
  - KEMRI CRDR Siaya Clinical Research Annex, Country Referral Hospital, Siaya, Siaya County
  - International Cancer Institute (ICI), Eldoret, Uasin Gishu County
  - Ahero Clinical Trials Unit, Kisumu
- Lebanon (2):
  - American University of Beirut Medical Centre, Hamra
  - Hospital Nini, Tripoli
- Netherlands (4):
  - Amsterdam UMC Lokatie VUMC, Amsterdam
  - Erasmus MC, Rotterdam
  - Haga Ziekenhuis, The Hague
  - UMC Utrecht, Van Creveldkliniek, Utrecht
- Nigeria (4):
  - University of Nigeria Teaching Hospital (UNTH), Ituku-Ozalla, Enugu State
  - Centre of Excellence for Sickle Cell Disease Research and Training, University of Abuja (CESRTA), Abuja, Federal Capital Territory (fct)
  - University College Hospital Paediatric Haematology and Oncology Unit, Ibadan, Ibadan, Oyo State
  - Lagos University Teaching Hospital, Lagos, Lagos
- Oman (2):
  - Sultan Qaboos University Hospital, Muscat, Sultanet of Oman/Muscat/Al Khoud
  - The Royal Hospital, Muscat
- Saudi Arabia (3):
  - King Abdulaziz Hospital-Al Ahsa-National Guard, Al Ahsa
  - National Guard Hospital Dammam, Dhahran
  - King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (8):
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Başkent Üniversitesi Adana-Hematoloji, Adana
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Hematoloji, Adana
  - Hacettepe University Hematology, Ankara
  - Hacettepe Üniversitesi Hastanesi- Hematoloji, Ankara
  - Mersin University Medical Faculty Pediatric Hematology, Mersin
  - Mersin Üniversitesi Tip Fakültesi Hastanesi- Çiftlikköy Yerleşkesi- Hematoloji, Mersin
  - VM Medical Park Mersin Hastanesi- Kardiyoloji, Mersin
- Uganda (3):
  - Makerere University College of Health Sciences (MakCHS), Kampala, Central Region
  - Joint Clinical Research Centre (JCRC), Kampala, Central Region (Wakiso District)
  - Jinja Regional Referral Hospital, Jinja, Eastern Region
- United Kingdom (6):
  - Addenbrooke's Hospital - Haemophilia and Thrombophilia, Cambridge
  - Whittington Hospital, London
  - Guy's Hospital - Haematology, London
  - King's College Hospital - Paediatric Research, London
  - Kings College Hospital - Haematology, London
  - Imperial College London, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com